CLINICAL TRIAL: NCT03824067
Title: Evaluation of the Impact of Point-of-Care Early Infant Diagnostic (EID) Testing on Timely Receipt of EID Results and Treatment Initiation in HIV-Exposed Children in Kenya and Zimbabwe
Brief Title: Impact of Point-of-Care EID for HIV-Exposed Infants
Acronym: POC-EID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EG0170
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2019-12

CONDITIONS: HIV/AIDS; Infant Morbidity; Pediatric HIV Infection; Transmission, Perinatal Infection
Keywords: HIV/AIDS; Point of Care; Early infant diagnosis; Health systems; Diagnostic tools; LMIC
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The design of this study is a cluster-randomized stepped wedge trial. This is whereby an intervention is rolled out sequentially to the study facilities over a number of time periods. The order in which the different clusters receive the intervention is determined at random and by the end of random allocation, all facilities will have received the intervention. Testing sites (determined from the list of all project facilities excluding pilot sites) will be randomized regarding timing of POC implementation; sites that serve as "hub" sites and their associated "spoke" sites will be given the same designation. The study will use a mixed method approach in data collection, and a qualitative component will also be conducted, including interviews and focus groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Early Infant Diagnosis (Active Comparator): Conventional laboratory based (standard of care - SOC) early infant diagnosis (EID) testing: SOC EID
  Interventions: Diagnostic Test: Standard of Care Early Infant Diagnosis
- Point of Care Early Infant Diagnosis (Experimental): The intervention is Point of Care (POC) early infant diagnosis (EID) testing, where the blood sample is processed at either the facility itself or a nearby site that is closer to the facility than a laboratory. With POC EID, blood samples do not have to travel to the laboratory for processing.
  Interventions: Diagnostic Test: Point of Care Early Infant Diagnosis

INTERVENTIONS:
Diagnostic Test: Point of Care Early Infant Diagnosis — HIV testing where the blood sample is processed at either the facility itself or a nearby site that is closer to the facility than a laboratory. With POC EID, blood samples do not have to travel to the laboratory for processing.
  Other Names: POC EID
  Arms: Point of Care Early Infant Diagnosis
Diagnostic Test: Standard of Care Early Infant Diagnosis — Conventional laboratory based EID testing
  Other Names: SOC EID
  Arms: Standard of Care Early Infant Diagnosis

SUMMARY:
This mixed methods study will utilize a randomized step-wedge design to assess the impact of point-of-care (POC) versus conventional early infant diagnosis (EID) on key outcomes including timely return of results to caregivers and time to initiation on treatment for HIV-infected infants. Data will be collected through longitudinal clinical follow-up and medical chart extraction of routine records and lab forms. Feasibility and acceptability data will be collected through interviews with mothers/caregivers of HIV-exposed infants, and community focus groups.

DETAILED DESCRIPTION:
This study seeks to evaluate the impact of point of care (POC) early infant HIV diagnosis (EID) on turn-around time from sample collection until notification of parents/caregivers of test result, linkage to care, and time to initiation of treatment, and early retention in HIV care (3-6 months) for those infected.

The study will take place in two countries, Zimbabwe and Kenya, with high HIV prevalence, and where EGPAF-supported POC EID platforms are being implemented as part of a Unitaid-funded POC EID project. As part of POC program implementation activities, in each country up to 50 EGPAF-supported sites will implement POC EID platforms. These sites may be prevention of mother-to-child transmission (PMTCT) of HIV clinics, HIV clinics or multidisciplinary health facilities. Project sites have been selected as part of the program implementation. In each country, 18 sites will be randomly selected as study sites for the impact evaluation.

Using a stepped wedge design, the intervention (the POC EID platforms) will be rolled out sequentially to the study facilities over three randomly-assigned time periods. Quantitative data will be derived from routine medical and laboratory charts and longitudinal tracking and follow-up of HIV-infected infants.

Qualitative data on feasibility and acceptability of POC will be derived from in-depth interviews with mothers/caregivers of HIV-exposed infants at the beginning and end of the study and community focus group discussions at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Any infant who receives an EID test, either conventional or POC, for the 4-6 week EID indication at one of the study sites (which were randomly selected from project sites in country)
* HEI under 12 weeks of age or their parents/caregivers
* Some methods will only include HEI who test positive (medical chart extraction and longitudinal follow up)
* Purposively selected caregivers of HEI for in-depth interviews
* Focus groups with community members will not require participants to have sought testing for EID

Exclusion Criteria:

* Participants not at selected study sites
* For some methods (medical chart extraction and longitudinal follow-up), HEI who test negative
* For qualitative component, excluded if unable to consent due to age, competence, or inability to speak any of the study languages

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9539 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of HIV exposed infants (HEI) who have received the 4-6 week EID test result by 12 weeks | 12 weeks
  The number of children for whom a sample was drawn for the 4-6-week indication receiving EID result by 12 weeks, divided by the number of HEI who presented to the clinic and had an indication for 4-6 week EID testing

SECONDARY OUTCOMES:
Testing coverage for the 4-6 week indication | 18 months
  Number of EID samples collected for 4-6 week indication divided by the number of HEI who presented to the clinic and had an indication for 4-6 week EID testing
Time from sample collection for 4-6 week EID test indication to parent's/ caregiver notification | 18 months
  Date of sample collection to the date that results were given to care giver
Age of patient at test result notification for 4-6 week EID test indication | 18 months
  HEIs date of birth, date of sample collection and date of result notification to care giver
Time from test result received for 4-6 week EID test to initiation of ART, for HIV-infected infants | 18 months
  Date positive result received at facility to the date the result was communicated to mother and date of ART initiation
Percentage of HIV positive infants diagnosed during 4-6 week EID testing initiated on ART | 18 months
  Number of HIV-infected infants initiated on ART after 4-6 week EID test divided by the number of HIV-infected infants identified after 4-6 week EID test
Number of HIV-infected infants diagnosed at the 4-6 week EID with retention in care at 6 months | 24 months
  Total number of infants initiated on ART 6 months ago and number of active on ART at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emma Sacks, PhD, Principal Investigator — George Washington University School of Public Health; Collins Odhiambo, MD, Principal Investigator — Elizabeth Glaser Pediatric Aids Foundation - Kenya; Agnes Mahomva, MD, Principal Investigator — Elizabeth Glaser Pediatric Aids Foundation - Zimbabwe; Jennifer Cohn, MD MPH, Study Director — Elizabeth Glaser Pediatric AIDS Foundation
Locations (2):
- Elizabeth Glaser Pediatric AIDS Foundation, Nairobi, Kenya
- Elizabeth Glaser Pediatric AIDS Foundation, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No